CLINICAL TRIAL: NCT03005873
Title: A Phase IIa, Randomized, Double Blinded, Placebo Controlled, Dose Finding Study for Single Dose Administration of TLC599 in Patients With Osteoarthritis (OA) of Knee
Brief Title: Phase IIa, Randomized, Double Blinded, Placebo Controlled, Dose Finding Study for TLC599 in OA Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiwan Liposome Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TLC599A2003
Record Dates: First submitted 2016-12-12; First posted 2016-12-29 (Estimated); Results first posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis of the knee; TLC599; Dexamethasone; DSP
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TLC599 LD group (Experimental): 12 mg DSP with 100 µmol PL (1.0 mL)
  Interventions: Drug: TLC599 LD group
- TLC599 HD group (Experimental): 18 mg DSP with 150 µmol PL (1.5 mL)
  Interventions: Drug: TLC599 HD group
- Placebo group (Placebo Comparator): 1.5 mL normal saline
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: TLC599 LD group — Single dose via intra-articular injection
  Other Names: 12 mg DSP with 100 µmol PL (1.0 mL)
  Arms: TLC599 LD group
Drug: Normal Saline — Single dose via intra-articular injection
  Other Names: Placebo
  Arms: Placebo group
Drug: TLC599 HD group — Single dose via intra-articular injection
  Other Names: 18 mg DSP with 150 µmol PL (1.5 mL)
  Arms: TLC599 HD group

SUMMARY:
This trial is a Phase IIa, Randomized, Double blinded, Placebo controlled, Dose finding Study to investigate the safety and efficacy of TLC599 in subjects with osteoarthritis of the knee.

DETAILED DESCRIPTION:
Protocol No: TLC599A2003 Name of Finished Product: TLC599

Title of Study:

A Phase IIa, Randomized, Double blinded, Placebo controlled, Dose finding Study for Single dose Administration of TLC599 in Patients with Osteoarthritis (OA) of Knee.

Study duration:

The trial will last around 27 weeks including a 21-day screening period and a 24-week follow-up period.

ELIGIBILITY:
Main Inclusion Criteria:

1. Male or female patients, at least 50 years of age.
2. Documented diagnosis of OA of the knee for at least 6 months
3. The study knee has OA with Grade 2 to 3 severity based on the Kellgren Lawrence grades
4. Patients with patient related visual analogue scale (VAS) score of 5.0 to 9.0 at baseline.
5. Willing and able to comply with study procedures and provide written informed consent.

Main Exclusion Criteria:

1. Patients who received systemic corticosteroids within the last 30 days prior to dosing.
2. Patients who use prohibited medications within 7 days prior to study drug administration or any pain control medication including acetaminophen within 48 hours prior to study drug administration.
3. Patients who use prohibited medications other than acetaminophen and oral NSAIDs from screening visit to 7 days prior to study drug administration.
4. Documented history and confirmed autoimmune disease
5. History of post-traumatic knee arthritis, or evidence of intra articular bleeding of the study knee
6. History of infective arthritis
7. Unstable study knee joint
8. Use of IA corticosteroid, hyaluronic acid, or other IA injection in the study knee within 3 months prior to the screening visit.
9. A history of treated malignancy which is disease free for ≤ 5 years prior to the screening visit
10. Uncontrolled and unstable concurrent medical or psychiatric illness, that will jeopardize the safety of the patient
11. Use of any chemotherapeutic or systemic immunosuppressant agents for inflammatory diseases within 6 months prior to the screening visit.
12. Current use of anticoagulants, including warfarin, heparin, low molecular weight heparin, or dabigatran.
13. Abnormalities of laboratory parameters as described below will qualify for exclusion:

    * hemoglobin < 8 g/dL;
    * total white blood cell count < 4000/ µL;
    * serum bilirubin/ alanine aminotransferase/ aspartate aminotransferase > 2 times upper limit of normal (ULN) for the laboratory reference ranges;
    * serum creatinine > 2 times ULN for the laboratory reference range;
    * serum uric acid > ULN for the laboratory reference range;
    * prothrombin time/International Normalized Ratio > ULN for the laboratory reference range.
14. Contraindication to undergoing magnetic resonance imaging (MRI)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Shih, PhD, Study Director — Taiwan Liposome Company
Locations (13):
- Australia (5):
  - Genesis Research Services Pty Limited, Broadmeadow
  - Pendlebury Clinic Private Hospital, Cardiff
  - Footscray Hospital- Western Health, Footscray
  - Linear Clinical Research Limited, Nedlands
  - Royal North Shore Hospital, Sydney
- Taiwan (8):
  - Show Chwan Memorial Hospital, Changhua
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Chung Shan Medical University Hosptial, Taichung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Cheng Hsin General Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Taipei Medical Universtiy Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hunter DJ, Chang CC, Wei JC, Lin HY, Brown C, Tai TT, Wu CF, Chuang WC, Shih SF. TLC599 in patients with osteoarthritis of the knee: a phase IIa, randomized, placebo-controlled, dose-finding study. Arthritis Res Ther. 2022 Feb 21;24(1):52. doi: 10.1186/s13075-022-02739-4. PMID 35189943

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TLC599 LD Group | TLC599 HD Group | Placebo Group
Started | 26 | 24 | 26
Completed | 25 | 21 | 22
Not Completed | 1 | 3 | 4
Not completed — Prohibited medication use post radnomization | 1 | 1 | 1
Not completed — Withdrew consent | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Ineligible post randomization | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: One patient from the Placebo group was enrolled but withdrawn from the analysis population due to ineligibility.
Groups:
- Total: Total of all reporting groups
Arm/Group | TLC599 LD Group | TLC599 HD Group | Placebo Group | Total
Number analyzed (Participants) | 26 | 24 | 25 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (9.07) | 62.9 (8.80) | 64.8 (8.45) | 63.9 (8.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 18 | 50
  Male | 11 | 7 | 7 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 22 | 24 | 72
  Unknown or Not Reported | 0 | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 13 | 13 | 12 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 13 | 11 | 13 | 37
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 13 | 12 | 12 | 37
  Australia | 13 | 12 | 13 | 38
VAS score (Study Knee) [Mean (Standard Deviation); unit: units on a scale] — The scores of the visual analog scale (VAS) are recorded by making a handwritten mark on a 10-cm line (from 0-cm to 10-cm) that represents a continuum between "no pain (0-cm)" and "worst pain (10-cm)". This is measured in millimeter from the left anchor "no pain (0-cm)" to generate a pain score.
  units on a scale | 6.45 (1.113) | 6.87 (1.215) | 6.56 (1.049) | 6.62 (1.125)
WOMAC Pain score (0-4) [Mean (Standard Deviation); unit: units on a scale] — The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain subscale consist of five items, each ranging from 0 to 4, making the total Pain subscore 0 to 20. The total score of the pain subscale for each patient is normalized and expressed on a 0 to 4 scale.
  Higher scores represent higher levels of pain (worse outcome), whereas lower scores represent lower levels of pain (better outcome).
  units on a scale | 1.49 (0.558) | 1.74 (0.631) | 1.62 (0.609) | 1.62 (0.600)
WOMAC Function score (0-4) [Mean (Standard Deviation); unit: units on a scale] — The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Function subscale consists of 17 items, each ranging from 0 to 4, making the total Function subscore 0 to 68. The total score of the Function subscale for each patient is normalized and expressed on a 0 to 4 scale.
  Higher scores represent higher levels of difficulty performing daily activities (worse outcome), whereas lower scores represent lower levels of difficulty performing daily activities (better outcome).
  units on a scale | 1.53 (0.531) | 1.82 (0.742) | 1.48 (0.652) | 1.61 (0.653)
Kellgren-Lawrence grades [Count of Participants; unit: Participants] — Kellgren-Lawrence (K-L) grading system is a method of classifying the severity of knee osteoarthritis (OA) using 5 grades:
  Grade 0: No radiographic features of OA are present; Grade 1: Doubtful joint space narrowing (JSN) and possible osteophytic lipping; Grade 2: Definite osteophytes and possible JSN on posteroanterior weight-bearing radiograph; Grade 3: Multiple osteophytes, definite JSN, sclerosis, possible bony deformity; Grade 4: Large osteophytes, marked JSN, severe sclerosis and definite bony deformity.
  Participants
    Grade 0 | 0 | 0 | 0 | 0
    Grade 1 | 0 | 0 | 0 | 0
    Grade 2 | 13 | 9 | 9 | 31
    Grade 3 | 13 | 15 | 16 | 44
    Grade 4 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in WOMAC Pain Subscale at Week 12
Description: The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain subscale consist of five items, each ranging from 0 to 4, making the total Pain subscore 0 to 20. The total score of the pain subscale for each patient is normalized and expressed on a 0 to 4 scale.
  Higher scores represent higher levels of pain (worse outcome), whereas lower scores represent lower levels of pain (better outcome).
  Missing data were imputed.
Time Frame: Baseline, Week 12
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | TLC599 LD Group | TLC599 HD Group | Placebo Group
Number analyzed (Participants) | 26 | 24 | 25
score on a scale | -0.83 (0.090) | -0.64 (0.094) | -0.47 (0.092)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | TLC599 LD Group | TLC599 HD Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 18/26 | 20/24 | 17/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TLC599 LD Group (N=26) | TLC599 HD Group (N=24) | Placebo Group (N=25)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TLC599 LD Group (N=26) | TLC599 HD Group (N=24) | Placebo Group (N=25)
Nasopharyngitis (Infections and infestations) | 4 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 4 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 2 | 0 | 1
Fungal skin infection (Infections and infestations) | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 6 | 4
Paraesthesia (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0
Piriformis syndrome (Nervous system disorders) | 0 | 0 | 1
Tension headache (Nervous system disorders) | 1 | 0 | 0
Cortisol decreased (Investigations) | 2 | 6 | 0
Lipase increased (Investigations) | 0 | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood calcium increased (Investigations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1
Heart rate irregular (Investigations) | 0 | 1 | 0
Hepatitis C virus test positive (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
White blood cells urine positive (Investigations) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 2
Joint injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Glucocorticoid deficiency (Endocrine disorders) | 3 | 1 | 0
Feeling hot (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0
Mass (General disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 2
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin lesion removal (Surgical and medical procedures) | 0 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT03005873/Prot_SAP_000.pdf